CLINICAL TRIAL: NCT05270161
Title: Comparative Evaluation of the Tunnel Technique and Free Gingival Graft in Gingival Recessions Treatment: Randomized Controlled Trial
Brief Title: The Tunnel Technique and Free Gingival Graft in Gingival Recessions Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Alfenas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFAlfenas
Record Dates: First submitted 2022-01-31; First posted 2022-03-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Esthetics; Gingiva
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Test Group 1 (T1) (Experimental): Multiple gingival recessions in the anterior region of the mandible treated with the tunnel technique.
  Interventions: Procedure: Tunnel technique; Procedure: Gingival graft - donor area
- Test Group 2 (T2) (Experimental): Isolate gingival recessions in the anterior region of the mandible treated with the laterally closed tunnel technique.
  Interventions: Procedure: Laterally closed tunnel technique; Procedure: Gingival graft - donor area
- Control Group 1 (C1) (Active Comparator): Multiple gingival recessions in the anterior region of the mandible will be treated using the free gingival graft technique.
  Interventions: Procedure: Free gingival graft; Procedure: Gingival graft - donor area
- Control Group 2 (C2) (Active Comparator): Isolate gingival recessions in the anterior region of the mandible will be treated using the free gingival graft technique.
  Interventions: Procedure: Free gingival graft; Procedure: Gingival graft - donor area
- Gel Group (G) (Experimental): The donor area on the palate will be treated using hyaluronic acid gel and green tea applied by the participant 3 times a day for 7 days.
  Interventions: Procedure: Gingival graft - donor area
- Clot Group (CO) (Active Comparator): No material will be placed in the donor area, only the clot will be kept in position by means of sutures.
  Interventions: Procedure: Gingival graft - donor area

INTERVENTIONS:
Procedure: Tunnel technique — Intrasulcular incisions on the buccal surface were made using a n°15 C blade, preserving the integrity of the papillae. The incision was extended to the adjacent tooth on both sides of the multiple recessions. Dissection of the entire buccal aspect was performed as a partial-thickness flap using sharp tunnel elevators preserving the papillae. The flap was extended beyond the mucogingival junction and under each papilla allowing a tension-free flap mobilization in the coronal direction. The connective tissue graft was placed in the tunnel and was stabilized using absorbable suspensory sutures. The mobilized mucous flap was advanced coronally to the cemento enamel junction, and suspensory sutures were stitched.
  Arms: Test Group 1 (T1)
Procedure: Laterally closed tunnel technique — Intrasulcular incisions on the buccal surface were made using a n°15 C blade, preserving the integrity of the papillae. The tunnel elevators were mobilized apically beyond the mucogingival line and extended medially and distally from the recession defect by undermining the facial surface of the interdental papillae. The insertion of muscles and fibers must be removed until a tension-free flap is obtained in the mesial, apical and distal directions. The preparation of the flap will be done carefully to avoid rupture of the papillae and perforation of the flap. As a result of this procedure, the mesial and distal margins of the flap must be brought together without tension to cover the exposed part of the root surface. The connective tissue graft was placed in the tunnel and was fixed mesially and distally at the inner aspect of the flap. Margins of the flap were pulled together over the graft and sutured with interrupted sutures.
  Arms: Test Group 2 (T2)
Procedure: Free gingival graft — In the recipient area, a marginal horizontal linear incision will be made in the mucogingival junction with a n°15 C blade, creating a partial thickness flap, keeping the periosteum intact. The horizontal dimension of the receiving area will be determined according to the mesiodistal extension of the area without keratinized gingiva. All mobile soft tissues, including epithelium, connective tissue and muscle fibers will be removed from the donor area using scissors to ensure stability in the recipient area. The connective tissue graft will be obtained by the free gingival graft technique and will be sutured in the recipient area.
  Arms: Control Group 1 (C1); Control Group 2 (C2)
Procedure: Gingival graft - donor area — The connective tissue graft will be obtained by the free gingival graft technique for all groups (T1, T2, T3 and T4). The mold of the prepared receiving area will be performed using sterile aluminum foil. The mold will be transferred to the donor area on the palate and the edges of the mold delimited with a scalpel blade. Deeper incisions will be made on the edges with the scalpel perpendicular to the palate, aiming to obtain a graft approximately 1.5 mm thick. With the scalpel blade parallel, the graft will be removed (epithelium and connective graft) maintaining its uniform thickness. For T1 and T2, the free gingival graft will be de-epithelialized. In donor area, a hyaluronic acid gel and green tea will be applied by the participant 3 times a day for 7 days (gel group) or no material will be placed in the donor area and the clot will be kept in position by means of sutures (clot group).

SUMMARY:
The present study aims to compare the tunnel technique/laterally closed tunnel technique and the FGG technique in the treatment of isolate/multiple GR in the anterior region of the mandible. Furthermore, it is proposed to evaluate the effect of a gel based on hyaluronic acid and green tea on the healing of the donor area after the removal of FGG from the palate. This work is expected to contribute to the still uncertain literature on the effectiveness of the tunnel technique as an alternative to the use of FGG in the treatment of multiple GR in the mandible.

DETAILED DESCRIPTION:
Free gingival graft (FGG) is a simple technique considered the most effective procedure to obtain gingival augmentation in sites with a minimal amount of keratinized gingiva. However, the abscence of chromatic integration and unsatisfactory texture of the graft after healing prevent its use in areas with high aesthetic demand. In this context, the tunnel technique (multiple gingival recessions [GR]) and the laterally closed tunnel technique (isolated GRs in the mandible) have been proposed as an alternative to the use of FGG in the treatment of GRs in the mandible. The present study aims to compare the tunnel technique/laterally closed tunnel technique and the FGG technique in the treatment of isolate/multiple GR in the anterior region of the mandible. Furthermore, it is proposed to evaluate the effect of a gel based on hyaluronic acid and green tea on the healing of the donor area after the removal of FGG from the palate. Sixty participants presenting isolate/multiple Miller Class I, II, or III GR [Recession type (RT) 1 or RT2] in the anterior region of the mandible will be included in the present study. Regarding the treatment of GR, participants will be divided into four groups: (1) Test Group 1 (T1) (n=15): multiple GR in the anterior region of the mandible treated with the tunnel technique; (2) Test Group 2 (T2) (n=15): isolate GR in the anterior region of the mandible treated with the laterally closed tunnel technique; (3) Control Group 1 (C1) (n=15): multiple GRs in the anterior region of the mandible will be treated using the FGG technique and (4) Control Group 2 (C2) (n=15): isolate GRs in the anterior region of the mandible will be treated using the FGG technique. Regarding the treatment of the donor area, the same participants will be divided into two groups: (1) Gel Group (G) (n=30): the donor area on the palate will be treated using hyaluronic acid gel and green tea applied by the participant 3 times a day for 7 days; (2) Clot Group (CO) (n=30): No material will be placed in the donor area, only the clot will be kept in position by means of sutures. Periodontal clinical parameters will be evaluated in the receiving area at the beginning of the study and after 1, 3, 6 and 12 months postoperatively. In the donor area, the percentage of wound closure, the epithelialized surface area and the color of the palatine mucosa will be evaluated in both groups after 3, 7, 15 and 30 days. The visual analogue scale (VAS) of pain (donor and recipient area) and aesthetic (recipient area) will be used to assess the participant's perception of the treatment used.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;
* Present isolated (≥4mm) or multiple GR in the anterior region of the mandible (tooth 33 to 43) Miller Class I, II or III (87) (or Recession type (RT) 1 or RT2);
* Systemically healthy with no contraindications for periodontal surgery;
* Probing depth of less than 3mm at the sites involved;
* Selected teeth properly positioned, free from endodontic treatment, any type of restorative treatment, caries or non-carious cervical lesion

Exclusion Criteria:

* Participants who use tobacco or other types of drugs;
* Participants submitted to periodontal treatment in the last 6 months;
* Pregnant participants;
* Participants who did not accept to return to follow-ups;
* Participants who used antibiotics, corticosteroids, chemotherapy, immunomodulators or others that modify the periodontal therapy results during the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
Recession depth | Change from baseline recession depth at 1, 3, 6 and 12 months
  Distance between cemento-enamel junction to free gingival margin.

SECONDARY OUTCOMES:
Recession width | Change from baseline recession width at 1, 3, 6 and 12 months
  Mesio-distal extent of gingival recession
Probing depth | Change from baseline probing depth at 1, 3, 6 and 12 months
  Distance between free gingival margin to the bottom of the sulcus.
Clinical attachment level | Change from baseline clinical attachment level at 1, 3, 6 and 12 months
  Distance between cemento-enamel junction to the bottom of the sulcus.
Keratinized tissue width | Change from baseline keratinized tissue width at 1, 3, 6 and 12 months
  Distance between the most apical point on free gingival margin to the mucogingival junction.
Gingival thickness | Change from baseline gingival thickness at 6 and 12 months
  The measurements were registered at the mid-buccal aspect of the tooth using a endodontic file. The distance between the marker and the tip of the file will be determined using a digital caliper.
Gingival margin position | Change from baseline gingival margin position at 1, 3, 6 and 12 months
  Distance from a reference point performed on the customized stent to the gingival margin.
Graft thickness after removal | Baseline
  Graft thickness will be assessed immediately after removal using a endodontic file in the middle of the graft. The distance between the marker and the tip of the file will be determined using a digital caliper.
Graft thickness immediately before suture | Baseline
  The thickness of the graft immediately before suturing will be evaluated after de-epithelialization (in the T group) and the removal of adipose tissue when present in both groups in the middle of the graft. The distance between the marker and the tip of the file will be determined using a digital caliper.
Height of keratinized tissue in graft | Change from immediate postoperative height of keratinized tissue in graft at 1, 3, 6 and 12 months
  Apico-coronal dimension of the graft measured at the stent mark using the periodontal probe.
Width of keratinized tissue in graft | Change from immediate postoperative width of keratinized tissue in graft at 1, 3, 6 and 12 months
  Mesio-distal dimension of the graft in the most coronal portion of the graft using the periodontal probe.
Graft contraction | Change from immediate postoperative graft contraction at 1, 3, 6 and 12 months
  Graft areas will be calculated by multiplying the height and width of keratinized tissue in graft.
Percentage of wound reduction by photographic image | Change from 3 days percentage of wound reduction by photographic image at 7, 15 and 30 days
  The millimeter periodontal probe will be positioned next to the wound at the time of obtaining the photos to calibrate the image analysis software that will be used to calculate the total area of the wound in donor region.
Percentage of Wound Reduction by clinical measurement | Change from 3 days percentage of wound reduction by clinical measurement at 7, 15 and 30 days
  The height and width of the wound will be determined using the periodontal probe.
Epithelized surface area | Change from 3 days epithelized surface area at 7, 15 and 30 days
  The epithelialization analysis will be performed using 3% oxygen peroxide to observe the presence of blistering in the wound. The absence of epithelialization will be characterized as blistering after contact of oxygen peroxide with the wound. This parameter will be noted dichotomously (presence/absence of bubbles), being noted as yes or no, respectively, in the participant's form.
Palatal mucosa color | Change from 3 days palatal mucosa color at 7, 15 and 30 days
  The color of the palatal mucosa will be evaluated by the visual analogue scale (VAS) in comparison with the color of the adjacent and opposite mucosa. In this evaluation, on a horizontal scale, 0 points will represent lack of color correspondence, 50 points will represent average correspondence and 100 points will represent excellent color correspondence with the adjacent tissues.
Postoperative complications | 3 days
  Presence of bleeding, swelling, infection and necrosis in the donor area will be recorded
Postoperative complications | 7 days
  Presence of bleeding, swelling, infection and necrosis in the donor area will be recorded
Landry index | Change from 3 days landry index at 7 and 30 days
  Classify the degree of repair based on erythema, presence of granulation tissue, bleeding/suppuration, and epithelialization in the recipient area. A score of 1 to 5 is given, where 1 is associated with a very poor/inadequate repair process and 5 is excellent.
Root coverage esthetic score (RES) | 6 months
  The RES system evaluates five variables of the recipient area including: gingival margin level, marginal tissue contour, soft tissue texture, JMG alignment and gingival color. Zero, 3 or 6 points will be used to assess the position of the gingival margin, while a score of 0 or 1 point will be used for each of the other variables. The ideal aesthetic score will be 10.
Root coverage esthetic score (RES) | 12 months
  The RES system evaluates five variables of the recipient area including: gingival margin level, marginal tissue contour, soft tissue texture, JMG alignment and gingival color. Zero, 3 or 6 points will be used to assess the position of the gingival margin, while a score of 0 or 1 point will be used for each of the other variables. The ideal aesthetic score will be 10.
Visual Analogue Scale (VAS) for pain | Change from 3 days VAS scale for pain at 7, 12 and 30 days
  The perception of pain will be recorded using the VAS scale at the operated sites. Participants will record the level of pain in the recipient and donor areas after the procedure on a horizontal scale, where the left endpoint will mean no pain (0), the midpoint of mean pain (50 ) and the right outcome severe pain (100).
Presence or absence of dentin sensitivity | Change from 1 month dentin sensitivity at 3, 6 and 12 months
  Determined from the participants' responses regarding the presence or absence of sensitivity in the cervical sites. For this, it will be asked if the participant has or not dentin sensitivity after a cold or air stimulus.
Visual Analogue Scale (VAS) for esthetics | 6 months
  Participants will be asked to express their overall satisfaction with treatment outcomes on a VAS scale, where the left endpoint will mean not at all satisfied (0), the midpoint reasonably satisfied (50) and the right endpoint extremely satisfied. satisfied (100).
Visual Analogue Scale (VAS) for esthetics | 12 months
  Participants will be asked to express their overall satisfaction with treatment outcomes on a VAS scale, where the left endpoint will mean not at all satisfied (0), the midpoint reasonably satisfied (50) and the right endpoint extremely satisfied. satisfied (100).
Analgesics consumption | 7 days
  The consumption of analgesics by the participants in the first 7 postoperative days will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suzane C Pigossi, PhD, Principal Investigator — Alfenas Federal University
Locations (1):
- Universidade Federal de Alfenas, Alfenas, Minas Gerais, Brazil

REFERENCES:
- [Derived] Oliveira JA, da Silveira MI, de Oliveira Alves R, Bezerra FJB, de Oliveira GJPL, Pigossi SC. Effect of a gel containing green tea extract and hyaluronic acid on palate pain scores and wound healing after free gingival graft: a quasi-randomized controlled clinical trial. Clin Oral Investig. 2023 Nov;27(11):6735-6746. doi: 10.1007/s00784-023-05282-x. Epub 2023 Sep 29. PMID 37775584